CLINICAL TRIAL: NCT04101708
Title: A Comparison of High-dose Dual Therapy and Half-dose Clarithromycin-containing Bismuth Quadruple Therapy for H.P Eradication in Elderly Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, director of Qilu Hospital gastroenterology department, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019SDU-QILU-G099
Record Dates: First submitted 2019-09-23; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Helicobacter Pylori
Keywords: elderly,helicobacter pylori eradication,dual therapy,half-dose clarithromycin
MeSH Terms: interventions — Lansoprazole; Amoxicillin; Clarithromycin; bismuth tripotassium dicitrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high dose dual group (Experimental): Patients in high dose dual group will receive lansoprazole (Takepron) 30mg po qid, amoxicillin 750mg po qid for 14d
  Interventions: Drug: Lansoprazole, Amoxicillin
- half-dose clarithromycin-containing bismuth quadruple group (Active Comparator): Patients in half-dose clarithromycin-containing bismuth quadruple group will receive lansoprazole (Takepron) 30mg po bid, amoxicillin 1000mg po bid, bismuth subcitrate (Colloidal Bismuth Pectin) 200mg po bid, and clarithromycin (Klacid) 250mg po bid for 14d
  Interventions: Drug: Lansoprazole, Amoxicillin,Clarithromycin and Bismuth subcitrate

INTERVENTIONS:
Drug: Lansoprazole, Amoxicillin — high dose dual regimen
  Arms: high dose dual group
Drug: Lansoprazole, Amoxicillin,Clarithromycin and Bismuth subcitrate — half-dose clarithromycin-containing bismuth quadruple regimen
  Arms: half-dose clarithromycin-containing bismuth quadruple group

SUMMARY:
The purpose of this study is to assess and compare the effectiveness and safety of high-dose dual therapy and half-dose clarithromycin-containing bismuth quadruple therapy in elderly patients for eradicating H.pylori.

DETAILED DESCRIPTION:
Helicobacter pylori plays an important role in many diseases such as peptic ulcer disease and MALT lymphomas. And the prevalence of H. pylori remains high in developing countries,including China.

Clarithromycin-containing bismuth quadruple therapy has been recommended as the first-line therapy for H pylori infection in China. However, its expensive cost and high antibiotic-related adverse reactions are always haunting us. In 2018,a research from NanFang hospital(China）revealed that 250mg clarithromycin is as effective as 500mg clarithromycin，at the same time，causes less adverse reactions. On the othe hand,previous studies reported a new regimen called large dose dual therapy（generally contains a PPI and amoxicillin),while some of them have achieved very good results,especially in Taiwan.

However, specific data on anti-H.pylori treatments in elderly people are very lacking.So,we aim to assess and compare the effectiveness and tolerability of high-dose dual therapy and half-dose clarithromycin-containing bismuth quadruple therapy in elderly patients.Considering the difference of drug metabolism between eldery and young people，a satisfactory result may be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Patients, aged greater than 65 , with positive H. pylori infection that was not eradicated by previous therapies are included. The H. pylori infection is confirmed by the positive rapid urease test or 13C-breath test.

Exclusion Criteria:

* Patients with significant underlying disease including liver, cardiac, pulmonary, and renal diseases, neoplasia, coagulopathy and genetic diseases, history of gastric surgery, pregnancy, breast-feeding, active gastrointestinal bleeding, the use of PPI, NSAID or antibiotics during the 4 weeks prior to enrolment, and previous history of allergic reactions to any of the medications used in this protocol. Patients previously treated with H. pylori eradication regimens or those unwilling to participate in the study were also excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-20 (Estimated); Primary Completion 2021-09-20 (Estimated); Study Completion 2022-09-20 (Estimated)

PRIMARY OUTCOMES:
eradication rate of the two groups | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, MD,PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu hosipital, Jinan, Shandong, China